CLINICAL TRIAL: NCT01485224
Title: Efficacy of Thalidomide in the Treatment of Severe Recurrent Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Efficacy of Thalidomide in the Treatment of Hereditary Hemorrhagic Telangiectasia
Acronym: THALI-HHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carlo Balduini, Professor of Internal Medicine, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudratCT 2011-004096-36
Record Dates: First submitted 2011-11-28; First posted 2011-12-05 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis
Keywords: Hereditary hemorrhagic telangiectasia; Epistaxis; Thalidomide
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide (Experimental): Single arm study:
  Eligible patients will receive thalidomide at a starting dose of 50 mg/day by mouth at bedtime for 4 weeks. In the event of unsatisfactory/no response, thalidomide dosage will be progressively increased by 50 mg/day every 4 weeks until complete or partial response, to a maximum dose of 200 mg/day.
  Treatment will be continued until one of the following criteria is met:
  * 8 additional weeks of treatment after the achievement of complete response
  * 16 additional weeks of treatment after the achievement of partial response
  * 24 weeks of treatment completed without response
  * unacceptable toxicity. Then, patients will be followed off of thalidomide for 24 weeks.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Eligible patients will receive thalidomide at a starting dose of 50 mg/day by mouth at bedtime for 4 weeks. In the event of unsatisfactory/no response, thalidomide dosage will be progressively increased by 50 mg/day every 4 weeks until complete or partial response, to a maximum dose of 200 mg/day.
  Treatment will be continued until one of the following criteria is met:
  * 8 additional weeks of treatment after the achievement of complete response
  * 16 additional weeks of treatment after the achievement of partial response
  * 24 weeks of treatment completed without response
  * unacceptable toxicity. Then, patients will be followed off of thalidomide for 24 weeks.
  Other Names: Thalidomide Celgene

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT) (OMIM 187300 and 600376), also known as Rendu-Osler-Weber syndrome, is an autosomal dominant disease and has a prevalence between 1:5000 and 1:8000 in different populations. Clinically, the occurrence of mucocutaneous and gastrointestinal telangiectasias and of systemic arteriovenous malformations is commonly observed. Recurrent and severe epistaxis, due to the presence of telangiectasias in nasal mucosa, is the most common presentation of HHT, frequently leading to severe anemia requiring intravenous iron and blood transfusions. Although not life threatening, severe epistaxis has a great impact on quality of life in HHT patients and it represents the most important impediment in daily activities, that poses therapeutic challenge. Recently, angiogenesis has been implicated in the pathogenesis of HHT. Circulating concentrations of both TGF-beta and vascular endothelial growth factor (VEGF) are significantly elevated and therefore, anti-angiogenic substances may be effective in the treatment of vascular malformations in this disease. Thalidomide functions as a potent immunosuppressive and antiangiogenic agent. The aim of this study is to assess the clinical effects of thalidomide therapy on the severity of epistaxis in subjects with HHT who are refractory to standard therapies.

DETAILED DESCRIPTION:
In the management of HHT epistaxis, multiple approaches have been tried, including electrocautery, laser, embolization, arterial ligation, but all approaches are largely palliative with variable results, many requiring repeated interventions. Except for nasal closure, surgical options offer, at best, limited hemorrhage-free intervals, but no definitive results and all have side effects. Moreover, currently, there is no established medical treatment available for these patients. To limit blood loss, the few medical treatments used include manipulation of the coagulation and fibrinolytic pathways or topical applications of anti-inflammatory drugs. However, multiple lesions disseminated over the entire mucosal surface are common in affected individuals, making local treatment difficult. Re-bleeding consumes a disproportionate share of healthcare resources devoted to multiple admissions, repeated endoscopies and blood transfusions.

Recently, angiogenesis has been implicated in the pathogenesis of HHT. Circulating concentrations of both TGF-beta and vascular endothelial growth factor (VEGF) are significantly elevated and therefore, anti-angiogenic substances may be effective in the treatment of vascular malformations in this disease.

Thalidomide functions as a potent immunosuppressive and antiangiogenic agent by inhibiting the phagocytic ability of inflammatory cells and the production of cytokines, such as tumor necrosis factor-alpha (TNF-a). It has been shown to be effective in the treatment of inflammatory diseases, in conditions associated with human immunodeficiency virus (HIV) infection, and in various cancers. Bleeding inhibition has been observed in HHT patients who received thalidomide as an antiangiogenic cancer therapy. A recent paper has reported that thalidomide treatment induced vessel maturation in an experimental model of HHT and reduced severe nosebleeds in six of the seven HHT patients studied. On the other hand, spectacular improvements have been described in patients with intestinal angiodysplasias, treated with thalidomide. In isolated case reports, patients with severe recurrent intestinal bleeding refractory to standard treatment achieved prolonged complete remission with thalidomide at a dose of 100 to 300 mg/day for a few months and tolerance was good. Cessation of bleeding was associated with a reduction in serum VEGF levels. These observations suggest that thalidomide might be useful for treatment of HHT patients and address significant unmet medical needs. Unfortunately, this drug exposes patients to the risk of severe side effects.

Drug metabolism is under control of a number of enzymes specific for each drug; among these enzymes, many show variable levels of activity and we can thus recognize in the population extensive (high or fast) metabolizers (EM) intermediate (IM) and poor (low or slow) metabolizers (PM). This is true also for thalidomide, whose metabolism is in part controlled by the enzyme CYP2C19.

The aims of our study are to test the hypothesis that thalidomide reduces the bleeding tendency of HHT patients and to verify to which extent CYP2C19 polymorphism modulates both response to treatment and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HHT, according to the diagnostic criteria world-wide recognized (Curacao criteria), with severe recurrent epistaxis (grade 2-3 according to the criteria proposed by Pagella et al., i.e. at least one episode of overt bleeding/week requiring at least one blood transfusion during the last three months), and refractory to mini-invasive surgical procedures, i.e. argon plasma coagulation. For these patients, there is no effective treatment option currently available
* Age > 18 years
* Ability of signing written informed consent
* Women of childbearing potential:
* declared intention not to start a pregnancy throughout the study and for four weeks following the date of the last dose of thalidomide (safe contraception, see Celgene guidelines, "Programma di Prevenzione della Gravidanza")
* negative serum pregnancy test obtained within 48 hours prior to the first dose of Thalidomide
* declared intention to undergo pregnancy tests periodically while on the study medication
* Males with female partner of childbearing potential:
* declared intention not to father throughout the study and for one week following the date of the last dose of thalidomide (safe contraception, see Celgene guidelines, "Programma di Prevenzione della Gravidanza")
* Estimated life expectancy must be greater than 10 months

Exclusion Criteria:

* Pregnant or lactating women, or potentially fertile (both males and females) who have not agreed to avoid pregnancy during the trial period and for four weeks (females) or one week (males) following the date of the last dose of thalidomide
* Neurological diseases
* Psychiatric illness that would prevent granting of informed consent
* Active cardiovascular disease
* High risk for thromboembolic events (comorbidities, such as diabetes or uncontrolled infections, malignancy, immobility, prior history of thromboembolic events, use of erythropoietic agents or other agents such as hormone replacement therapy, central venous catheter, anti-cardiolipin, or anti-beta2 glycoprotein antibodies)
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption since thalidomide capsules contain lactose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2016-10-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients showing a decrease in the frequency, intensity and duration of epistaxis and in the blood transfusion requirement. | up to 24 weeks
  Cessation of nose bleeding will be defined as complete response. Reduction in the severity of any bleeding parameter less than complete response will represent partial response.

SECONDARY OUTCOMES:
Size and number of telangiectasias evaluated by endoscopy of nasal mucosa (recording images of the size and localization of telangiectasias) | up to 24 weeks
Minimum dose of the drug that reduces bleeding | up to 24 weeks
Time to response | up to 24 weeks
Time to relapse after the end of treatment | up to 24 weeks after the end of treatment
Number of adverse events | up to 1 year
Correlations between biological parameters, response to treatment and side effects profile | up to 24 weeks
  * Correlations between the mutations that are responsible for HHT and response to treatment
  * Correlations between polymorphisms of CYP2C19 and response to treatment
  * Correlations between polymorphisms of CYP2C19 and side effects profile

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Balduini, M.D., Principal Investigator — Fondazione IRCCS Policlinico S. Matteo, Pavia, Italy
Locations (1):
- Clinica Medica 3, Fondazione IRCCS Policlinico S. Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebrin F, Srun S, Raymond K, Martin S, van den Brink S, Freitas C, Breant C, Mathivet T, Larrivee B, Thomas JL, Arthur HM, Westermann CJ, Disch F, Mager JJ, Snijder RJ, Eichmann A, Mummery CL. Thalidomide stimulates vessel maturation and reduces epistaxis in individuals with hereditary hemorrhagic telangiectasia. Nat Med. 2010 Apr;16(4):420-8. doi: 10.1038/nm.2131. Epub 2010 Apr 4. PMID 20364125
- [Derived] Invernizzi R, Quaglia F, Klersy C, Pagella F, Ornati F, Chu F, Matti E, Spinozzi G, Plumitallo S, Grignani P, Olivieri C, Bastia R, Bellistri F, Danesino C, Benazzo M, Balduini CL. Efficacy and safety of thalidomide for the treatment of severe recurrent epistaxis in hereditary haemorrhagic telangiectasia: results of a non-randomised, single-centre, phase 2 study. Lancet Haematol. 2015 Nov;2(11):e465-73. doi: 10.1016/S2352-3026(15)00195-7. Epub 2015 Oct 27. PMID 26686256